CLINICAL TRIAL: NCT06670807
Title: Clinical Trial to Evaluate the Efficacy of a Probiotic Formula on Cognitive Function in Mild Cognitive Impairement Patients.
Brief Title: Effect of a Probiotic Formula in Mild Cognitive Impairement
Acronym: PROBIOMIND
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: AB Biotics, SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CPP2022-009632
Record Dates: First submitted 2024-10-23; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Mild Cognitive Impairment (MCI)
Keywords: Mild Cognitive Impairment (MCI); Probiotic; Cognitive function; Microbiota; Nutrition; Elderly
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Active Comparator): Probiotic formulation that includes L. plantarum CECT 7481, L. plantarum CECT 7485 Y L. brevis CECT7480
  Interventions: Dietary Supplement: Probiotic Arm
- Control Group (Placebo Comparator): Placebo comparator arm with identical pharmaceutical form and aspect, containing microcrystalline cellulose
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic Arm — Fifty of the participants will consume 1 capsule/day of the dietary supplement AB-MIND+CECT7481 for 16 weeks. The capsule should be taken just before breakfast. The researchers will instruct the volunteers to maintain their usual lifestyle (diet, physical activity, sleep habits) throughout the intervention period.
  Other Names: AB-MIND+CECT7481
  Arms: Experimental group
Other: Placebo — Fifty of the participants will consume 1 capsule/day of the PLACEBO for 16 weeks. The capsule should be taken just before breakfast. The researchers will instruct the volunteers to maintain their usual lifestyle (diet, physical activity, sleep habits) throughout the entire intervention period.
  Arms: Control Group

SUMMARY:
Mild cognitive impairment is currently one of the most relevant social challenges, as its prevalence is expected to increase and it is associated with a higher risk of developing Alzheimer's disease or other types of dementia. Therefore, it is necessary to seek strategies that can be applied in the early stages to delay or reverse the progression of the disease.

In this context, probiotics have emerged as a promising alternative for managing cognitive disorders. This project is a clinical-nutritional trial to evaluate the utility of consuming a dietary supplement containing probiotics on the cognitive function of individuals with mild cognitive impairment. The study will involve 100 participants, selected from the Geriatrics Unit of San Carlos Clinical Hospital, as well as through various Leisure Centers in Madrid, randomly assigned to two groups of 50 individuals each (Experimental Group and Control Group). Participants assigned to the experimental group will consume the dietary supplement, while those in the control group will receive a placebo, which is a product without probiotics. Both groups will take 1 capsule per day of the assigned product at breakfast for 16 weeks. During this time, changes will be analyzed in various imaging tests, cognitive tests, and some blood parameters related to cognitive function. Changes in gut microbiota and different lifestyle factors (diet, body composition, physical activity, sleep) will also be evaluated.

DETAILED DESCRIPTION:
Currently, the number of Alzheimer's disease (AD) cases is reaching epidemic proportions. In the European Union, the prevalence of Alzheimer's disease increases from 2% in individuals aged 65-69 to 22% in those aged 85-89, and this figure is expected to double due to the demographic aging of the population by 2040, placing an unprecedented burden on society (Jané-Llopis & Gabilondo, 2008). These statistics highlight the urgent need for intervention strategies that counteract the progression of the disease, particularly in the early stages of mild cognitive impairment (MCI), and delay the onset of the most debilitating clinical symptoms.

As is well known, the etiopathophysiology of cognitive decline is multifactorial, involving both non-modifiable factors (e.g., sex, genetics) and modifiable ones (e.g., lifestyle). Among the latter are poor-quality diets, physical inactivity, smoking, and altered sleep patterns, which directly impact key risk factors for cognitive decline, such as hypertension, hypercholesterolemia, and obesity. Moreover, recent studies have observed that diet and other lifestyle factors seem to significantly influence the composition of the gut microbiota, which in turn may directly affect the gut-brain axis and the pathogenesis of dementias (Kesika et al., 2021). This opens the door to new therapeutic options based on microbiota-modifying strategies.

In this context, probiotics have emerged as a promising alternative for the management of cognitive disorders due to their ability to beneficially modulate the gut microbiota and, consequently, the gut-brain axis. However, it is important to note that probiotic properties are strain-specific, meaning that a given strain must be thoroughly investigated before such properties can be ascribed (Hill et al., 2014).

Three probiotic strains, in particular, have shown potential positive effects on gut-brain axis modulation and intestinal barrier reinforcement in previous studies, mainly in vitro. These strains are **L. brevis** CECT 7480, **L. plantarum** CECT 7485, and **L. plantarum** CECT 7481 (L. plantarum DR7™). Specifically:

* L. brevis CECT 7480 has demonstrated a high capacity for GABA production in in vitro experimental studies, as well as broad antagonism against opportunistic pathogens (Bosch et al., 2012; Ferrés-Amat et al., 2020).
* L. plantarum CECT 7485 appears to improve intestinal permeability and modulate the gut-brain axis through increased acetylcholine (ACh) production and has shown antagonism against opportunistic intestinal pathogens (Perez et al., 2020).
* Additionally, L. plantarum CECT 7485 and L. brevis CECT 7480 have recently been investigated in two clinical trials related to stress, anxiety, and depression, showing beneficial effects (Denysov et al., 2023). However, to date, these strains have not been studied in other pathologies affecting the central nervous system (CNS) and cognition, such as MCI in aging populations.
* L. plantarum CECT 7481 (L. plantarum DR7™) has shown, in both in vitro studies and clinical trials, positive neuromodulatory effects through the regulation of enzymes involved in neurotransmitter pathways such as serotonin, kynurenine, and norepinephrine. Metabolomic analyses have also demonstrated that it increases ACh levels. Furthermore, significantly lower plasma cortisol levels (Chong et al., 2019) and reductions in oxidative stress and plasma peroxidation (Chong et al., 2019a) were detected following L. plantarum D administration in adults. Changes in gut-brain axis pathways correlated with modifications in the gut bacterial composition in adults (Liu et al., 2020). Clinical evidence showed a positive impact of L. plantarum DR7 on stress and anxiety, as well as improved cognitive function as a secondary outcome. However, these findings were evaluated in healthy adults, and its use in MCI patients requires a specific clinical trial to validate its effects.

Considering the importance of neurotransmitter circuits involved in MCI and AD (Solas et al., 2015), this clinical trial hypothesizes that the administration of a dietary supplement containing the combination of the three aforementioned probiotic strains could have great potential to improve cognitive function by reinforcing the intestinal barrier, preventing gut dysbiosis, and, most importantly, modulating the gut-brain axis.

The clinical trial will be divided into two phases: the Selection Phase and the Experimental Phase.

Selection Phase Additionally, the three strains meet safety prerequisites (verified in vitro, in vivo, and in clinical studies) and have QPS (Qualified Presumption of Safety) status from EFSA, which, if positive results are found in the clinical study, would facilitate the future commercialization of a dietary supplement aimed at populations with MCI to help prevent the progression of cognitive decline.

Individuals interested in participating in the study, who have previously been informed about its characteristics at the Geriatrics Unit of the Hospital Clínico San Carlos and the associated Community Centers (Moncloa and Chamartín), will be invited to the Faculty of Pharmacy at the Complutense University of Madrid (Visit 0, V0) to assess eligibility criteria through:

* Medical history: A semi-structured clinical interview focusing on health-related data to verify the fulfillment of selection criteria, including family history, medical treatments, neurological/psychiatric diseases, and other conditions (e.g., cancer), history of alcoholism, etc.
* Cognitive and functional assessment questionnaires to verify the selection criteria: MoCA (Nasreddine et al., 2005), CDR (Morris, 1993), and (I)ADL.

Once eligibility is confirmed, participants will be given a patient information sheet providing detailed information on the study's design and features. The principal investigator will also provide a verbal summary of the study. After addressing any questions and ensuring understanding, those interested in participating will sign the informed consent form.

Additionally, participants may also choose to provide informed consent for storing leftover biological samples in the National Biobank Registry, in accordance with Royal Decree 1716/2011, as outlined in the informed consent form.

Once informed consents are signed, participants will receive the following questionnaires and materials to complete and return at their next visit (V1):

* Dietary Study Questionnaires (Food Frequency Questionnaire, Adherence to the Mediterranean Diet)
* Container and instructions for stool collection
* Accelerometers and instructions

At the end of V0, appointments will be scheduled for the various tests to be performed at the initial visit (V1), all to be completed within a maximum period of 7 days:

* Appointment for blood analysis
* Appointment for MRI
* Appointment for magnetoencephalographyand neuropsychological tests
* Appointment for the lifestyle study, including the collection of questionnaires and materials provided at V0, and the provision of guidelines.

EXPERIMENTAL PHASE

Following the selection visit (V0), participants will begin the 16-week intervention period of the experimental phase of the study. During this period, they will attend the following visits:

Visit 1 (V1 (initial visit of the intervention period)

During this visit, researchers will collect a series of variables for the following studies (described in section 7.2.4):

* COGNITIVE FUNCTION STUDY (Faculty of Psychology, UCM): The research team's psychologists will collect data related to cognitive function:
* Magnetoencephalography/EEG and MRI will be performed.
* In addition to the tests completed in V0 (MoCA and CDR), the following tests will be conducted:
* Cognitive reserve assessment
* Typical cognitive function tests
* Functional capacity tests
* Psychiatric symptom tests
* Assessment of subjective perceptions of memory, language, and executive function decline
* Psychosocial parameter tests
* BLOOD ANALYSIS (Partner Laboratory): A fasting blood sample (minimum of 8 hours) will be collected to determine relevant biochemical parameters.
* MICROBIOTA STUDY(Faculty of Pharmacy, UCM): Stool samples will be collected to determine gut microbiota composition.
* LIFESTYLE STUDY (Faculty of Pharmacy, UCM): Researchers will perform the following:
* Dietary study: Review questionnaires submitted during V0 (Food Frequency Questionnaire, Adherence to the Mediterranean Diet). The first 24-hour dietary recall will be conducted, and participants will be informed that this questionnaire will be repeated two more times via phone within a week.
* Anthropometric study: Body measurements and composition will be recorded.
* Physical activity study: Physical activity will be assessed using a validated questionnaire and accelerometry.
* Sleep habits study: Sleep quality and chronotype will be evaluated using specific questionnaires and accelerometry.
* Other health indicators: Quality of life and vital signs will be measured.

After collecting the variables from these studies, the researchers will provide the participants with instructions according to the randomization list. Specifically, participants will be instructed to take one capsule per day of the assigned product with breakfast for the next 16 weeks. They will also be advised to maintain their usual diet and lifestyle (physical activity, sleep) during this period. The necessary supply of capsules will be provided to last until the final visit.

Finally, participants will receive questionnaires and materials to complete and return at the final visit (V5):

* Dietary Study Questionnaires (Food Frequency Questionnaire, Adherence to the Mediterranean Diet)
* Container and instructions for stool collection
* Accelerometers and instructions
* Treatment adherence and tolerance control sheet
* Adverse effects control sheet

The date for the final visit will be confirmed in follow-up phone calls and reminders sent one week in advance by phone or message, emphasizing the need to bring the completed materials from V1.

V2 (Week 4); V3 (Week 8); V4 (Week 12)

Telephone follow-up interviews will be conducted, including:

* Evaluation of adherence and tolerance to the product
* Recording of adverse events

Visit 5 (V5) (Week 16) (Final visit of the intervention period):

During this visit, the researchers will collect the same variables taken during the initial visit (V1) and will also administer the MoCA and CDR tests that were conducted during V0 to complete the cognitive function assessment at the end of the intervention period.

Additionally, the following will be carried out:

* Assessment of adherence and tolerance to the product consumption
* Recording of adverse events

A database will be created in Excel, equipped with a double-entry system and filters to prevent and detect any inconsistencies or errors. The information will be cleaned and validated. Descriptive analysis will be conducted for qualitative data (absolute frequencies, percentages) and quantitative data (mean, standard deviation, median, interquartile range, minimum, and maximum). Differences between groups will be analyzed using Chi-square tests, and quantitative data will be analyzed with the appropriate test based on the distribution of the variables.

The data will be analyzed in a blinded manner by the principal investigator of the study, in collaboration with the Research Support Unit of the Information Technology and Technical User Support Area at Complutense University of Madrid. Statistical analysis will be performed using SPSS version 29.0 (SPSS Inc.) or later versions..

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 60 and 85 years.
* Present "Mild Cognitive Impairment" (MCI) based on:
* MoCA test (< 26 points) or score adjusted for educational level
* and CDR test (≤ 0.5 points)
* Maintain functional capacity according to the (I)ADL test (≥ 70 points)
* Show "cognitive concern" reported by the participant and/or a surrogate caregiver
* Demonstrate longitudinal decline in cognitive function (progressive and not stabilized) for more than 3-5 years.
* BMI ≥ 20 and < 30 kg/m²
* Absence of a family or social environment that prevents treatment adherence.
* Adequate cultural level and understanding of the clinical study.
* Agree to participate voluntarily in the study and provide written informed consent.

Exclusion Criteria:

* Subjects with severe neurological or psychiatric disorders due to any of the following causes: severe dementia, depression, epilepsy, schizophrenia, or bipolar disorder.
* Subjects who have suffered a severe stroke prior to the study (FAZKAS=3)
* Subjects with a history of malignancy < 5 years (< 5 years if the brain was affected)
* Subjects who have experienced severe traumatic brain injury with structural brain injury and/or prior brain surgery
* Subjects with pacemakers and those with metal implants that may interfere with EEG or MRI
* Subjects treated with medications: benzodiazepines, neuroleptics, narcotics, anticonvulsants, or sedative-hypnotics in the last 3 months
* Subjects who have been treated with antibiotics or probiotic supplements at least 3 months before the start of the study.
* Subjects with hearing or visual impairments that prevent the evaluations included in the study
* Subjects with severe illnesses affecting nutritional status (liver, kidney, etc.)
* Subjects who have engaged in weight loss diets or significant dietary changes in the 8 weeks prior to starting the study
* Subjects with high alcohol consumption (> 3 alcoholic beverages per day)

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in cognitive function by electrophysiological study | From enrollment to the end of treatment at 16 weeks
  Changes in cognitive function evaluated by studying variations in the functional network through phase hypersynchrony in the alpha band, measured using an electrophysiological study.
  Functional network of the brain will be recorded using an Electroencephalography (EEG) with 128 channels. 20 minutes of resting state activity will be recorded for each participant: 10 minutes with opened eyes and 10 minutes with closed eyes. The signal will be filtered in-line between 0.1 and 300 Hz, sampled at a sampling rate of 1000 Hz. The recordings will be preprocessed using the spatio-temporal filtering algorithm tSSS (Taulu, 2009) with the software Maxfilter software (supplied by Elekta) to remove magnetic noise and compensate for head movements during the recordings.

SECONDARY OUTCOMES:
Change in global cognitive function by MoCA test | From enrollment to the end of treatment at 16 weeks
  Changes in global cognitive function will be analyzed by Montreal Cognitive Assessment test (MoCA) before the intervention, and at the end of the treatment at 16 weeks. The score range of MoCA is 0-30.
Change in global cognitive function by CDR test | From enrollment to the end of treatment at 16 weeks
  Changes in global cognitive function will be analyzed by Clinical Dementia Rating (CDR) before the intervention, and at the end of the treatment at 16 weeks. The CDR is based on a scale of 0-3: no dementia (CDR = 0), questionable dementia (CDR = 0.5), MCI (CDR = 1), moderate cognitive impairment (CDR = 2), and severe cognitive impairment (CDR = 3).
Change in verbal episodic memory by WMS-III | From enrollment to the end of treatment at 16 weeks
  Changes in verbal episodic memory will be analyzed by Wechsler Memory Scale 3rd edition (WMS-III) before the intervention, and at the end of the treatment at 16 weeks. The WMS-III has most representative standardization databases to assess memory and make optimal clinical recommendations. The 11 subtests that comprise the index scores average 60 min, ranging from 45 to 75 min, to administer. The time needed to administer the 13 subtests required to generate all of the summary and index scores is 80 min, with a range of 65 to 95 min.
Change in verbal fluency by Boston Naming Test | From enrollment to the end of treatment at 16 weeks
  Changes in verbal fluecy will be analyzed by Boston Naming Test (BNT) before the intervention, and at the end of the treatment at 16 weeks. BNT measures word retrieval. The range is 0-60 with higher representing better performance.
Change in mood by Geriatric Depression Scale | From enrollment to the end of treatment at 16 weeks
  Changes in mood will be analyzed by a short version of the Geriatric Depression Scale (GDS). This test is a self-assessment scale often used in geriatric depression trials. The GDS is a 15-item screening tool used to identify depression in older adults. In scoring the Geriatric Depression Scale, each item is scored 0 or 1. The total score on the scale ranges from 0 to 15 with higher scores indicating worse outcome.
Change in Serum Brain Derived Neurotrophic Factor (BDNF) concentration | From enrollment to the end of treatment at 16 weeks
  Serum BDNF will be estimated by ELISA using human BDNF ELISA kit from Boster Biological Technology Co. Ltd., Pleasanton, CA. Higher levels of serum BDNF (ng/mL) are optimal.
Change in serum Gamma-Amino Butyric Acid (GABA) concentration | From enrollment to the end of treatment at 16 weeks
  Concentrations of GABA (ng/mL) will be measured in serum samples by LC-MS.
Change in plasma acetycholine level | From enrollment to the end of treatment at 16 weeks
  Plasma acetycholine concentration (nmol/L) will be measured using choline oxidase-mediated enzyme coupling reactions (AAT Bioques, Inc., Sunnyvale, CA, USA) according to the manufacturer's instructions.
Change in Tumour necrosis factor (TNF)-alpha, interleukin (IL) 6 and IL-10 levels | From enrollment to the end of treatment at 16 weeks
  The cytokines IL-6, IL-10 and TNF-alpha will be analyzed using the Enzyme-linked immunosorbent assay (ELISA) method and reported their levels in pg/ml.
Change in composition of gut microbiota | From enrollment to the end of treatment at 16 weeks
  Gut microbiota composition will be analyzed using 16s rRNA DNA sequencing method.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Facultad de Farmacia Universidad Complutense de Madrid (UCM) Plaza Ramón y Cajal, Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid, Madrid

IPD SHARING:
Plan to Share IPD: No
The tested product may lead to a patent